CLINICAL TRIAL: NCT04788030
Title: Outcome After Reconstruction of 43 Digital Nerve Lesions With Muscle-in-Vein Conduits
Brief Title: Reconstruction of Digital Nerve Lesions With Muscle-in-Vein Conduits
Status: Completed | Type: Observational
Sponsor: BG Trauma Center Tuebingen (Other)
Responsible Party: Principal Investigator, PD Dr. Theodora Wahler, Chief of the Department of Hand, Plastic and Aesthetic Surgery, medius Hospital Nürtingen, BG Trauma Center Tuebingen
Other Study IDs: 650/2018BO2-1
Record Dates: First submitted 2021-02-19; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Peripheral Nerve Injury Upper Limb

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Digital nerve reconstruction with muscle-in-vein conduits
  Interventions: Other: Nerve reconstruction

INTERVENTIONS:
Other: Nerve reconstruction — Nerve bridging with muscle-in-vein conduits

SUMMARY:
Muscle-in-vein conduits (MVCs) provide an alternative for bridging digital nerve defects when tension-free suture is not possible. Low donor site morbidity and absence of additional costs are favorable advantages compared to autografts or conduits. 37 patients with 43 defects of proper palmar digital nerves were retrospectively enrolled. Primary repair by MVCs was performed in 22 cases while 21 underwent secondary reconstruction. Recovery of sensibility was assessed by static and moving two-point discrimination (2PDs, 2PDm) and Semmes-Weinstein monofilaments (SWM). Results were compared with contralateral side serving as intraindividual control. Outcome data were stratified according to international guidelines and evaluated for differences in terms of age, gap length, time of reconstruction and concomitant injuries.

ELIGIBILITY:
Inclusion Criteria:

- Patients with reconstruction of digital nerves with muscle-in-vein conduits

Exclusion Criteria:

* Subtotal or total amputations
* pre-existing neurological disorders (e.g. polyneuropathy)
* symptoms of nerve entrapment

Ages: 6 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The mean age of all patients was 38.0 years (SD 18.4, range 6-72). All patients aged younger than 18 years were males whereas patients older than 60 years tend to be females.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Two-point discrimination | Six months after reconstruction or later
Semmes-Weinstein-Monofilament test | Six months after reconstruction or later

SECONDARY OUTCOMES:
Age | Baseline
Gap length | Baseline
Time of reconstruction | Baseline
Concomitant injuries | Baseline

IPD SHARING:
Plan to Share IPD: Undecided